CLINICAL TRIAL: NCT02377505
Title: Deep Brain Stimulation in Treatment Resistant Schizophrenia: Randomized, Controlled, Crossover Pilot Study
Brief Title: Deep Brain Stimulation in Treatment Resistant Schizophrenia
Acronym: DBS-SCHIZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-ECP-2013-20; PI12/00042 (Other: Fundació Institut Recerca-Hospital Santa Creu i Sant Pau)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Refractory Schizophrenia
Keywords: Treatment-Resistant Schizophrenia; Deep Brain Stimulation
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-Stimulation (Active Comparator): Disease condition is assessed with stimulation turned "on"
  Interventions: Device: On-Stimulation
- Off-Stimulation (Placebo Comparator): Disease condition is assessed with stimulation turned "off"
  Interventions: Device: Off-Stimulation

INTERVENTIONS:
Device: On-Stimulation — The surgical electrode implanted in target 1 (mPFC) or target 2 (NAcc) by a pulse generating device (Kinetra, Medtronic Inc) is "on"
  Arms: On-Stimulation
Device: Off-Stimulation — The surgical electrode implanted in target 1 (mPFC) or target 2 (NAcc) by a pulse generating device (Kinetra, Medtronic Inc) is "off"
  Arms: Off-Stimulation

SUMMARY:
This study aims at assessing efficacy and safety of Deep Brain Stimulation (DBS) for treatment of patients with treatment resistant schizophrenia, by means of a random, controlled and crossed study.

DETAILED DESCRIPTION:
The first phase of the study will consist of implanting electrodes. Recruited patients will be random to 2 targets: (1) medial prefrontal cortex (mPFC); (2) nucleus accumbens (NAcc). Continuous stimulation will be applied until the patients stabilise clinically. This period is anticipated between 6 and 9 months.

After this stage, the next phase will consist of the crossover study. Those patients who respond to DBS will be randomly distributed in two groups, for a period of 3 months: on stimulation group and off stimulation group. Patients will then be crossed over to the other group for a further 3 months.

Weekly visits during first month after, and fortnightly visits will be made during the entire study to evaluate treatment efficacy and patient tolerance.

Patients who complete the study and respond to treatment with DBS will be provided continuing with treatment, and keeping control visits to assess the long-term effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 55 years.
2. DSM IV-TR diagnosis of schizophrenia for at least 3 years prior to the screening visit.
3. Determined to be treatment-resistant as demonstrated by:

   1. Persistence of positive symptoms which have not responded to appropriate treatments for at least 2 years.
   2. Inadequate response from adequate trials of two different classes of antipsychotic drugs (not including clozapine), at least 8 weeks.
   3. Inadequate response from adequate trial of clozapine, at least 3 months, or unable to tolerate clozapine because of intolerable side effects.
   4. ECT is contraindicated or have failed to produce a maintained response.
4. Persistence of positive symptoms defined as i) requiring a score of 4 (mild) or more on at least 2 of the next PANSS items: delusions, hallucinatory behavior, suspiciousness and unusual thought content; or as ii) requiring a score of 6 (severe) or more on at least 1 of the above PANSS items.
5. Current CGI score 6 or more
6. Stable antipsychotic treatment for last 2 months.
7. Women of childbearing age using medically approved contraceptive methods.
8. Adequate familiar or social support during all study procedures.

Exclusion Criteria:

1. MRI (Magnetic Resonance Imaging) contraindication to stimulation or contraindications for MRI
2. History of epilepsy or clozapine-induced seizures, where use of anticonvulsants was needed
3. Current suicidal ideation, plan or intent for self-harm during last 2 months.
4. Evidence of global cognitive impairment.
5. Current acute, serious or unstable illnesses.
6. History of substance abuse (other than tobacco or caffeine).
7. Comorbid axis I or II DSM IV-TR disorders.
8. Female patients who are pregnant or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Changes from baseline score to 1-3 weeks scores and to fortnightly scores until the end of trial (12 months)
  Scale to assess changes in schizophrenia' symptoms

SECONDARY OUTCOMES:
Clinical Global Impression-Schizophrenia (CGI-SCH) | Changes from baseline score to 1-12 months scores
  Scale to assess changes in schizophrenia symptoms' severity, global improvement or change.
Global Functioning Scale (GFS) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess changes in social, occupational, and psychological functioning
Social Functioning Scale (SFS) | Changes from baseline score to 1-3 weeks scores and to 1-12 months scores
  Scale to assess changes in social functioning
Personal and Social Performance (PSP) | Changes from baseline score to 1-12 months scores
  Scale to assess changes in functioning
Psychotic Symptom Rating Scales (PSYRATS) | Changes from baseline score to 1-12 months scores
  Scale to assess changes in hallucinations
Scale for the Assessment of Negative Symptoms (SANS) | Changes from baseline score to 1-12 months scores
  Scale to assess changes in negative symptoms of schizophrenia
Calgary Depression Scale for Schizophrenia (CDSS) | Changes from baseline score to 1-12 months scores
  Scale to assess changes in depressive symptoms
Performance-Based Skills Assessment (UPSA) | Changes from baseline score to 12 months score
  Scale to assess changes in functional capacity
Neuropsychological Assessment | Changes from baseline score to 12 months score
  Battery of neuropsychological tests to assess changes in cognition
Cerebral metabolism (PET scans) | Changes from baseline scan to 6 and 12 months scans
  Assessment of changes in brain blow flow using the nuclear medicine procedure, PET
n-Back (fMRI scan) | Changes from baseline scan to 6 and 12 months scans
  Task to measure changes in working memory
Adverse events (AEs) | Changes from baseline score to 1-3 weeks scores and to fortnightly scores until the end of trial (12 months)
  All unexpected medical problem that happens during DBS treatment

CONTACTS AND LOCATIONS:
Overall Officials: Iluminada Corripio, MD, PhD, Principal Investigator — Department of Psychiatry. Hospital Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - FIDMAG Germanes Hospitalàries Research Foundation, Sant Boi de Llobregat, Barcelona
  - Department of Psychiatry. Hospital Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salgado-Lopez L, Pomarol-Clotet E, Roldan A, Rodriguez R, Molet J, Sarro S, Alvarez E, Corripio I. Letter to the Editor: Deep brain stimulation for schizophrenia. J Neurosurg. 2016 Jul;125(1):229-30. doi: 10.3171/2015.12.JNS152874. Epub 2016 Apr 22. No abstract available. PMID 27104842
- [Result] Corripio I, Sarro S, McKenna PJ, Molet J, Alvarez E, Pomarol-Clotet E, Portella MJ. Clinical Improvement in a Treatment-Resistant Patient With Schizophrenia Treated With Deep Brain Stimulation. Biol Psychiatry. 2016 Oct 15;80(8):e69-70. doi: 10.1016/j.biopsych.2016.03.1049. Epub 2016 Mar 10. No abstract available. PMID 27113497
- [Result] Corripio I, Roldan A, Sarro S, McKenna PJ, Alonso-Solis A, Rabella M, Diaz A, Puigdemont D, Perez-Sola V, Alvarez E, Arevalo A, Padilla PP, Ruiz-Idiago JM, Rodriguez R, Molet J, Pomarol-Clotet E, Portella MJ. Deep brain stimulation in treatment resistant schizophrenia: A pilot randomized cross-over clinical trial. EBioMedicine. 2020 Jan;51:102568. doi: 10.1016/j.ebiom.2019.11.029. Epub 2020 Jan 8. PMID 31927311